CLINICAL TRIAL: NCT03956368
Title: A Randomised, Double-blind, Placebo-controlled Trial on the Efficacy of Atorvastatin in Chronic Subdural Haematoma (The REACH Study)
Brief Title: Efficacy of Atorvastatin in Chronic Subdural Haematoma
Acronym: REACH
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Wai Sang Poon, Chair Professor & Chief in Neurosurgery, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REACH-v1
Record Dates: First submitted 2019-05-10; First posted 2019-05-20 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Chronic Subdural Hematoma
Keywords: Chronic subdural haematoma; Medical treatment; Atorvastatin; Clinical outcome; Surgical recurrence
MeSH Terms: conditions — Hematoma, Subdural, Chronic | interventions — Atorvastatin

STUDY DESIGN:
Intervention Model Description: Eligible subjects will be randomised upon admission to receive atorvastin 20mg nocte or placebo for 8 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Randomised on the day of admission to receive oral Atorvastatin 20mg daily for 8 weeks.
  Interventions: Drug: Atorvastatin 20mg
- Control Group (Placebo Comparator): Randomised on the day of admission to receive placebo 20mg daily for 8 weeks.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Atorvastatin 20mg — 20mg (every evening orally) for 8 weeks.
  Arms: Treatment Group
Drug: Placebos — 20mg (every evening orally) for 8 weeks.
  Arms: Control Group

SUMMARY:
This prospective, double-blind, randomized, placebo-controlled study aims to evaluate the efficacy and safety of atorvastatin in patients with chronic subdural haematoma. The degree of disability or dependence in daily activities, as well as surgical intervention or recurrence, of the treatment and control groups will be compared.

DETAILED DESCRIPTION:
Objectives: Chronic subdural haematoma (CSDH) is a common neurosurgical condition in the elderly population associated with mild head injury. Surgical drainage has been regarded as safe and effective. However, surgical complications including recurrences can result in poor functional outcome and fatality, particularly in the elderly patients. Atorvastatin, an HMGCoA reductase inhibitor and a widely prescribed lipid lowering medication has properties of inflammation modulation and neovasculature promotion.

Hypothesis: Atorvastatin can improve functional outcome in patients with CSDH for both initially non-operatively treated group (estimated to be 10%) and the operative group (90%) by reducing the rate of surgical intervention and recurrence rate.

Design: A prospective multicentre study of 690 consented patients with symptomatic CSDH will be randomised on the day of admission to receive atorvastatin 20 mg or a placebo daily for 8 weeks. All seven regional neurosurgical units in Hong Kong and two units outside Hong Kong, each treating 80-200 patients per annum, have been invited to participate.

Main Outcome Measures: Primary outcome: Modified Rankin Scale (mRS). Secondary outcome: surgical recurrence.

Sample Size: Assuming an absolute 10% improvement in favourable outcome in the Modified Rankin Scale score (mRS 0-3) at 6 months from the control group of 70% to the treatment group 80%, allowing a 10% loss to follow up, a sample size of 690 is required.

Expected Results: A successful study for improving clinical outcome of CSDH, an important illness of the elderly with an annual incidence of 58/100,000 will change clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years old;
2. Evidence of supratentorial chronic subdural haematoma (unilateral or bilateral) by Computed Tomography (CT);
3. Patients are joining the trial voluntarily with consent form signed.

Exclusion Criteria:

1. Allergy to atorvastatin or other statins;
2. Deranged liver function;
3. Patients who are already on long term steroid for other condition(s);
4. Patients who are already on statin for other condition(s);
5. Presence of cerebrospinal fluid diversion device (e.g. ventriculo-peritoneal shunt);
6. Pregnant or on breast feeding;
7. Hematoma is secondary to tumour or haematological disorders;
8. Patients taking angiotensin converting enzyme (ACE) inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 690 (Estimated)
Dates: Start 2020-01-09 (Actual); Primary Completion 2022-09-16 (Estimated); Study Completion 2023-03-16 (Estimated)

PRIMARY OUTCOMES:
Favourable Modified Rankin Scale (mRS) score | 6 months
  Modified Rankin Scale score of 0-3

SECONDARY OUTCOMES:
Chronic subdural haematoma (CSDH) related surgical intervention | Throughout the study period, an average of 6 months
  Recurrence rate in both initially non-operatively treated patients and operative cases

OTHER OUTCOMES:
Glasgow Outcome Scale (GOS) | 2 weeks, 8 weeks, 3 months, and 6 months
  Gross clinical outcome measure which allows standardised descriptions (good recovery, moderate disability, severe disability, persistent vegetative state, and death, with good recovery indicating the best outcome and death indicating the worst) for the degree of recovery in patients with brain damage.
Imaging diagnosis | Index admission, 1-2 weeks early post-operation or before discharge, 3 months, 6 months
  Computed Tomography (CT) brain scan to exclude the presence of air and new blood in subdural space at 1-2 weeks and to elevate the clarification of CSDH resolution at 3 months and 6 months.
Barthel Index (BI) | 2 weeks, 8 weeks, 3 months, and 6 months
  Ordinal scale used to measure performance in activities of daily living (ADL) which uses 10 variables describing ADL and mobility. Scores range from 0-100 with 0 indicating the worst outcome and 100 indicating the best outcome.
Montreal Cognitive Assessment (MoCA) | 2 weeks, 8 weeks, 3 months, and 6 months
  One-page test for detecting cognitive impairment. The score ranges from 0-30 with a higher score indicating better outcome.
Modified Rankin Scale | 2 weeks, 8 weeks, 3 months, and 6 months
  Scale for measuring the degree of disability or dependence in the daily activities of patients with brain injury.

CONTACTS AND LOCATIONS:
Overall Officials: Wai Sang Poon, MBChB-Glasg FRCSEd FHKAM-Surg, Principal Investigator — Chinese University of Hong Kong
Locations (7):
- Hong Kong (7):
  - Prince of Wales Hospital, Shatin, New Territories
  - Pamela Youde Nethersole Eastern Hospital, Chai Wan
  - Queen Mary Hospital, Hong Kong
  - Kwong Wah Hospital, Kowloon
  - Princess Margaret Hospital, Kowloon
  - Queen Elizabeth Hospital, Kowloon
  - Tuen Mun Hospital, Tuenmen